CLINICAL TRIAL: NCT02532517
Title: A Prospective, Multi-center, Single Arm Study to Evaluate the Safety and Effectiveness of the CODMAN ENTERPRISE® Vascular Reconstruction Device and Delivery System When Used in Conjunction With Endovascular Coil Embolization in the Treatment of Wide-necked Saccular Intracranial Aneurysms
Brief Title: Study to Evaluate the Safety and Effectiveness of the CODMAN ENTERPRISE® Vascular Reconstruction Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No safety issues; change in innovation strategy
Sponsor: Cerenovus, Part of DePuy Synthes Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NV-IDE-1001
Record Dates: First submitted 2015-08-24; First posted 2015-08-25 (Estimated); Results first posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-09

CONDITIONS: Intracranial Aneurysm
Keywords: CODMAN ENTERPRISE® Vascular Reconstruction Device; Wide Neck, Intracranial, Saccular Aneurysms; Cerebral Aneurysms
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Enterprise (Experimental)
  Interventions: Device: CODMAN ENTERPRISE® Vascular Reconstruction Device and Delivery System

INTERVENTIONS:
Device: CODMAN ENTERPRISE® Vascular Reconstruction Device and Delivery System

SUMMARY:
The purpose of this study is to demonstrate effectiveness and safety of the CODMAN ENTERPRISE® Vascular Reconstruction Device and Delivery System.

DETAILED DESCRIPTION:
The study is a prospective, multi-center, single arm, clinical study to evaluate the safety and effectiveness of the ENTERPRISE stent when used in conjunction with endovascular coil embolization in the treatment of unruptured wide-neck, intracranial, saccular anterior circulation aneurysms (≤ 10 mm). The primary objectives of the study are to evaluate the rate of complete angiographic occlusion at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Target aneurysm is an unruptured wide-neck, intracranial, saccular anterior circulation aneurysm (≤ 10 mm) arising from a parent vessel with a diameter of ≥ 2.5 mm and ≤ 4 mm
* Subject understands the nature of the procedure and provides voluntary written informed consent prior to the treatment
* Subject is willing to comply with specified follow-up evaluation

Exclusion Criteria:

* Planned staged procedure
* Currently enrolled in another investigational device or drug study
* Target aneurysm that has been previously treated
* Mycotic, fusiform or dissecting aneurysm
* Admission platelet <50,000 or any known hemorrhagic diathesis, coagulation deficiency, or on oral anticoagulant therapy with an INR >3.0
* A serum creatinine level > 2.5 mg/dL within 7 days prior to index procedure

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Frei, MD, Principal Investigator — Radiology Imaging Associates
Locations (11):
- United States (11):
  - Radiology Imaging Associates, Englewood, Colorado
  - University of Florida, Gainesville, Florida
  - Lyerly Neurosurgery, an Affiliate of Baptist Health, Jacksonville, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - University of Buffalo, Buffalo, New York
  - Mount Sinai Health System, New York, New York
  - Miami Valley Hospital, Dayton, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Inova Fairfax Hospital, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- CODMAN ENTERPRISE: Participants with an unruptured wide-neck, intracranial saccular anterior circulation aneurysm (less than or equal to [<=] 10 millimeters [mm]), arising from a parent vessel with a diameter of greater than or equal to [>=] 2.5 mm and <= 4 mm, treated with either CODMAN ENTERPRISE Vascular Reconstruction Device and Delivery System (ENTERPRISE VRD system) and or CODMAN ENTERPRISE 2 Vascular Reconstruction Device and Delivery System (ENTERPRISE 2 VRD system).
Period: Overall Study
Arm/Group | CODMAN ENTERPRISE
Started | 45
mITT Analysis Set | 44
Completed | 28
Not Completed | 17
Not completed — Did not complete 24-Month visit | 4
Not completed — Failed Angiographic eligibility | 1
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 4
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-treat (mITT) analysis set is defined as participants who were found to be eligible for treatment of ENTEPRISE during pre-procedure angiographic assessment, and in whom treatment is attempted.
Arm/Group | CODMAN ENTERPRISE
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.4 (12.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 38
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Aneurysm Occlusion (RCAO) Without Retreatment at 12-Month Post Procedure
Description: The Raymond-Roy Grading scale used for judging intracranial aneurysm (IA) endosaccular embolization success ranges from Grade I to III where, Grade I is completion occlusion with no flow of contrast seen in the aneurysm sac, Grade II is partial occlusion with some flow or eddy flow in the aneurysm sac and Grade III is residual aneurysm or Incomplete occlusion with apparent flow in the aneurysm sac. RCAO was assessed by the Independent Core Laboratory, complete aneurysm occlusion is defined as an aneurysm in which a Grade I (completion occlusion), is achieved on the Raymond Scale at the relevant post-procedure angiogram, without additional procedures for treatment of the aneurysm since the index procedure. Participants who were retreated (retreatment includes staged procedures) prior to the 12-month were considered not to have achieved complete aneurysm occlusion.
Time Frame: 12 Months Post Procedure
Population: Modified Intent to Treat (mITT) analysis set: participants who were found to be eligible for treatment of ENTEPRISE during pre-procedure angiographic assessment, and in whom treatment is attempted. Here 'N' (Number of participants analyzed) included all participants available at 12-month visit with non missing values for this outcome measure (OM).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | CODMAN ENTERPRISE
Number analyzed (Participants) | 22
Percentage of Participants | 81.8 [59.7 to 94.8]

2. Primary Outcome: Percentage of Participants With Major Ipsilateral Stroke and/or Death Due to Ipsilateral Stroke at 12 Months Post Procedure
Description: The incidence of a major ipsilateral stroke and/or death due to ipsilateral stroke was evaluated from the start of the index procedure until completion of the 12-month follow-up. A major ipsilateral stroke is defined as a new neurological event which is ipsilateral and in the vascular distribution territory of the stenting procedure and that results in an increase of greater than or equal to (>=) 4 on the National Institute of Health Stroke Scale (NIHSS) as compared to baseline and persists for greater than 24 hours. The NIHSS is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. The scores range from 0 to 42 with a score of 0 indicates no stroke; 1-4 as minor stroke; 5-15 as moderate stroke; 15-20 as moderate/severe stroke; 21-42 as severe stroke. NIHSS worsening is defined as an increase from baseline of >= 4.
Time Frame: At 12 Months Post Procedure
Population: mITT analysis set defined as participants who were found to be eligible for treatment of ENTEPRISE during pre-procedure angiographic assessment, and in whom treatment is attempted. Here 'N' (Number of participants analyzed) signifies participants who have been followed-up to the timepoint of interest (12 months) in the population for this OM.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CODMAN ENTERPRISE
Number analyzed (Participants) | 40
Percentage of participants
  Ipsilateral Stroke | 7.5 [1.6 to 20.4]
  Death related to Ipsilateral Stroke | 0 [0.0 to 0.0]

3. Primary Outcome: Percentage of Participant With In-Stent Stenosis at 12 Months Post Procedure Per Independent Core Laboratory
Description: In-stent stenosis is defined as greater than 50 percent (%) narrowing of the vessel within the ENTERPRISE stent or within 10 millimeters (mm) of either end of the stent.
Time Frame: At 12 Months post procedure
Population: mITT analysis set is defined as participants who were found to be eligible for treatment of ENTEPRISE during pre-procedure angiographic assessment, and in whom treatment is attempted. Here 'N' (Number of participants analyzed) signifies all participants who were available at the 12-month visit with non-missing values for this OM.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CODMAN ENTERPRISE
Number analyzed (Participants) | 23
Percentage of participants | 0.0 [0.0 to 14.8]

4. Secondary Outcome: Number of Participants With Procedure Success Immediately Post-procedure (Acute), 6 and 12 Months
Description: The procedure success rate is defined to be the percentage of aneurysms in which coil mass position is maintained within the sac with parent artery patency, without additional procedures for treatment of the aneurysm since the index procedure. The procedure success was summarized immediately post-treatment (acute), and at the 6- and 12-month follow-up assessments.
Time Frame: Immediately post-procedure (acute), 6 and 12 months
Population: mITT analysis set is defined as participants who were found to be eligible for treatment of ENTEPRISE during pre-procedure angiographic assessment, and in whom treatment is attempted. Here 'n' (number analyzed) signifies participants available at specified visits with non-missing values of the OM.
Measure: Count of Participants; unit: Participants
Arm/Group | CODMAN ENTERPRISE
Number analyzed (Participants) | 44
Participants
  Immediately post-procedure (acute) | 41
  6-Month Follow-up: number analyzed (Participants) | 35
  6-Month Follow-up | 34
  12-Month Follow-up: number analyzed (Participants) | 23
  12-Month Follow-up | 23

5. Secondary Outcome: Number of Participants With Complete Aneurysm Occlusion as Per the Raymond Scale Immediately Post-procedure (Acute), 6 and 12 Months
Description: The Raymond-Roy Grading scale used for judging intracranial aneurysm (IA) endosaccular embolization success ranges from Grade I to III where, Grade I is completion occlusion with no flow of contrast seen in the aneurysm sac, Grade II is partial occlusion with some flow or eddy flow in the aneurysm sac and Grade III is residual aneurysm or Incomplete occlusion with apparent flow in the aneurysm sac. RCAO was assessed by the Independent Core Laboratory, complete aneurysm occlusion is defined as an aneurysm in which a Grade I (completion occlusion), is achieved on the Raymond Scale at the relevant post-procedure angiogram, without additional procedures for treatment of the aneurysm since the index procedure. Participants who are retreated (retreatment includes staged procedures) prior to the 12-month were considered not to have achieved complete aneurysm occlusion.
Time Frame: Immediately post-procedure (acute), 6 and 12 months
Population: mITT analysis set included. Here 'N' (Number of participants analyzed) signifies all evaluable participants with valid assessments post procedure for this OM and 'n' (number analyzed) signifies participants available at the schedule visits with non-missing values of the OM.
Measure: Count of Participants; unit: Participants
Arm/Group | CODMAN ENTERPRISE
Number analyzed (Participants) | 42
Participants
  Immediately post-procedure (acute) | 16
  6-Month Follow Up: number analyzed (Participants) | 34
  6-Month Follow Up | 24
  12-Month Follow Up: number analyzed (Participants) | 22
  12-Month Follow Up | 18

6. Secondary Outcome: Number of Participants With Complete/Partial Aneurysm Occlusion as Per the Raymond Scale Immediately Post-procedure (Acute), 6 and 12 Months
Description: The Raymond-Roy Grading scale used for judging intracranial aneurysm (IA) endosaccular embolization success ranges from Grade I to III where, Grade I is completion occlusion with no flow of contrast seen in the aneurysm sac, Grade II is partial occlusion with some flow or eddy flow in the aneurysm sac and Grade III is residual aneurysm or Incomplete occlusion with apparent flow in the aneurysm sac. Complete/partial aneurysm occlusion is defined as an aneurysm in which a score of 1 (complete occlusion) or 2 (residual neck) is achieved on the Raymond Scale, regardless of retreatment. Participants who are retreated (retreatment includes staged procedures) prior to the 12-month post-procedure follow-up visit was considered not to have achieved complete aneurysm occlusion.
Time Frame: Immediately post-procedure (acute), 6 and 12 Months
Population: mITT analysis set included. Here 'N' (Number of participants analyzed) signifies all evaluable participants with valid assessments post procedure for this OM and 'n' (number analyzed) signifies number of participants available at the specified visits with non-missing values of the OM.
Measure: Count of Participants; unit: Participants
Arm/Group | CODMAN ENTERPRISE
Number analyzed (Participants) | 42
Participants
  Immediately post-procedure (acute) | 34
  6-Month Follow Up: number analyzed (Participants) | 34
  6-Month Follow Up | 32
  12-Month Follow Up: number analyzed (Participants) | 22
  12-Month Follow Up | 21

7. Secondary Outcome: Number of Participants With 25% to 100% Aneurysm Occlusion Immediately Post-procedure (Acute), 6 and 12 Months
Description: Number of Participants with aneurysms occlusion of 100%, 90%-99%, 70-89%, 50-69%, 25-49%, or <25% occlusion in accordance with Consensus Grades 0 (100% complete aneurysm occlusion) - 5 (<25% volumetric aneurysm occlusion), respectively, was reported immediately post-procedure (acute), and at the 6 and 12 month follow-up, respectively.
Time Frame: Immediately post-procedure (acute), 6 and 12 months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | CODMAN ENTERPRISE
Number analyzed (Participants) | 42
Participants
  Immediately post-procedure (acute): 100% | 16
  Immediately post-procedure (acute): 90% - 99% | 26
  Immediately post-procedure (acute): 70% - 89% | 0
  Immediately post-procedure (acute): 50% - 69% | 0
  Immediately post-procedure (acute): 25% - 49% | 0
  Immediately post-procedure (acute): <25% | 0
  6-Month Follow-up: number analyzed (Participants) | 34
  6-Month Follow-up: 100% | 24
  6-Month Follow-up: 90% - 99% | 8
  6-Month Follow-up: 70% - 89% | 2
  6-Month Follow-up: 50% - 69% | 0
  6-Month Follow-up: 25% - 49% | 0
  6-Month Follow-up: <25% | 0
  12-Month Follow-up: number analyzed (Participants) | 22
  12-Month Follow-up: 100% | 18
  12-Month Follow-up: 90% - 99% | 3
  12-Month Follow-up: 70% - 89% | 1
  12-Month Follow-up: 50% - 69% | 0
  12-Month Follow-up: 25% - 49% | 0
  12-Month Follow-up: <25% | 0

8. Secondary Outcome: Number of Participants With Aneurysm Recanalization
Description: Number of participants with aneurysm recanalization was reported. Recanalization was defined as an increase in aneurysm filling as compared to the previous study-specified angiographic assessment, resulting in a change in (that is, worsening of) the Raymond classification.
Time Frame: Up to 12 months
Population: mITT analysis set is defined as participants who were found to be eligible for treatment of ENTEPRISE during pre-procedure angiographic assessment, and in whom treatment is attempted. Here 'N' (number of participants analyzed) included all evaluable participants with data available for this OM.
Measure: Count of Participants; unit: Participants
Arm/Group | CODMAN ENTERPRISE
Number analyzed (Participants) | 23
Participants | 2

9. Secondary Outcome: Number of Participants Retreated With Any Additional Treatment
Description: Retreatment was defined as any additional treatment of the target aneurysm after the index procedure (retreatment includes staged procedures), or an additional procedure (regardless of whether retreatment is by surgery or endovascular treatment) due to recanalization, rupture or bleeding.
Time Frame: Up to 12 months
Population: mITT analysis set: participants who were found to be eligible for treatment of ENTEPRISE during pre-procedure angiographic assessment, and in whom treatment is attempted. Here 'N' (number of participants analyzed) included participants who had been followed up to 12-month follow-up, or otherwise who were retreated prior to 12-Month Follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | CODMAN ENTERPRISE
Number analyzed (Participants) | 37
Participants | 0

10. Secondary Outcome: Number of Participants With New Neurological Deficits as Per the Modified Rankin Scale (mRS) Score
Description: Observed scores on the Modified Ranking Scale was presented at baseline (pre-procedure) and follow-up (30 days, 6 and 12 months post-procedure). mRS score: 0 = no symptoms at all; 1 = no significant disability despite symptoms, able to carry out all usual duties and activities; 2 = slight disability, unable to carry out all previous activities but able to look after own affairs without assistant; 3 = moderate disability, requires some help, but able to walk without assistance; 4 = moderate to severe disability, unable to walk without assistance, and unable to attend own bodily needs without assistance; 5 = severe disability, bedridden, incontinent, and requiring constant nursing care and attention; 6 = dead. The number of participants who had an increase in mRS > 2 from baseline not related to stroke or death was also be presented for each follow-up time point.
Time Frame: Post-procedure up to 30-Day, 6-Month Follow-up and 12-Month Follow-up
Population: mITT analysis set: participants who were found to be eligible for treatment of ENTEPRISE during pre-procedure angiographic assessment, and in whom treatment is attempted. Here 'n' (number analyzed) signifies number of participants available at the specified visits with non-missing values of the OM.
Measure: Count of Participants; unit: Participants
Arm/Group | CODMAN ENTERPRISE
Number analyzed (Participants) | 44
Participants
  Post-procedure up to 30-Day Follow-up | 5
  Post-procedure up to 6-Month Follow-up: number analyzed (Participants) | 43
  Post-procedure up to 6-Month Follow-up | 5
  Post-procedure up to 12-Month Follow-up: number analyzed (Participants) | 34
  Post-procedure up to 12-Month Follow-up | 5

11. Secondary Outcome: Number of Participants With NIH Stroke Scale (NIHSS) Worsening
Description: The National Institutes of Health Stroke Scale (NIHSS) is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. The scores range from 0 to 42 with a score of 0 indicates no stroke; 1-4 as minor stroke; 5-15 as moderate stroke; 15-20 as moderate/severe stroke; 21-42 as severe stroke. NIHSS worsening is defined as an increase from baseline of >= 4.
Time Frame: Post-procedure up to 6-Month and 12-Month Follow-up
Population: mITT analysis set included. Here 'N' (Number of participants analyzed) included participants who had at least one post-baseline NIHSS scores and 'n' (number analyzed) signifies number of participants analyzed at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | CODMAN ENTERPRISE
Number analyzed (Participants) | 38
Participants
  Post-procedure up to 6-Month Follow-up | 2
  Post-procedure up to 12-Month Follow-up: number analyzed (Participants) | 30
  Post-procedure up to 12-Month Follow-up | 2

12. Secondary Outcome: Number of Participants With Reduced Thrombolysis in Cerebral Infarction (TICI) Flow (New Occurrence of TICI Grade of 0 or 1)
Description: The percentage of target aneurysms in which a new occurrence of unintentional and persistent reduced TICI flow (TICI grade of 0: No perfusion or 1: Partial perfusion) was observed at the target vessel during the index procedure as a result of a mechanical obstruction such as dissection or luminal thrombus was evaluated. TICI evaluates perfusion severity and ranges from Grade 0 (No perfusion) to 3 (Complete perfusion).
Time Frame: Day 1 (Intraoperative)
Population: mITT analysis set is defined as participants who were found to be eligible for treatment of ENTEPRISE during pre-procedure angiographic assessment, and in whom treatment is attempted.
Measure: Count of Participants; unit: Participants
Arm/Group | CODMAN ENTERPRISE
Number analyzed (Participants) | 44
Participants | 2

13. Secondary Outcome: Number of Participants With Bleeding Complications
Description: The number of participants who experienced a procedure-related hemorrhagic event which required any of the following was evaluated: blood transfusion, surgical intervention, a new hospitalization, or lengthening of hospital stay. The complications of hematoma requiring treatment (that is, hematoma > 5 centimeter [cm] in diameter occurring at the access site) and retroperitoneal bleeding were reported as hemorrhagic events.
Time Frame: 12 months
Population: mITT analysis set included. Here 'N' (Number of participants analyzed) included all participants with data available for this OM and 'n' (number analyzed) signifies number of participants analyzed at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | CODMAN ENTERPRISE
Number analyzed (Participants) | 37
Participants
  Post-procedure up to 6-Month Follow-up | 3
  Post-procedure up to 12-Month Follow-up: number analyzed (Participants) | 26
  Post-procedure up to 12-Month Follow-up | 3

14. Secondary Outcome: Number of Participants With In-Stent Stenosis Per Independent Core Laboratory During Procedure (Acute), Post-procedure up to 6 Months and 12 Months Follow up
Description: In-stent stenosis is defined as greater than 50% narrowing of the vessel within the ENTERPRISE stent or within 10 mm of either end of the stent.
Time Frame: During procedure (acute), post-procedure up to 6 months and 12 months follow up
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | CODMAN ENTERPRISE
Number analyzed (Participants) | 42
Participants
  During procedure (acute) | 0
  Post-procedure up to 6-Month Follow-up: number analyzed (Participants) | 35
  Post-procedure up to 6-Month Follow-up | 0
  Post-procedure up to 12-Month Follow-up: number analyzed (Participants) | 23
  Post-procedure up to 12-Month Follow-up | 0

15. Secondary Outcome: Number of Participants With Thrombosis Per Independent Core Laboratory
Description: Thrombosis is defined as in-stent thrombosis.
Time Frame: During procedure (acute), post-procedure up to 6 months and 12 months follow up
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | CODMAN ENTERPRISE
Number analyzed (Participants) | 42
Participants
  During procedure (acute) | 1
  Post-procedure up to 6-Month Follow-up: number analyzed (Participants) | 35
  Post-procedure up to 6-Month Follow-up | 0
  Post-procedure up to 12-Month Follow-up: number analyzed (Participants) | 23
  Post-procedure up to 12-Month Follow-up | 0

ADVERSE EVENTS:
Time Frame: Up to 24 months
Description: mITT analysis set is defined as participants who were found to be eligible for treatment of ENTEPRISE during pre-procedure angiographic assessment, and in whom treatment is attempted.
Arm/Group | CODMAN ENTERPRISE
All-Cause Mortality (participants affected / at risk) | 4/44
Serious Adverse Events (participants affected / at risk) | 14/44
Other Adverse Events (participants affected / at risk) | 24/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CODMAN ENTERPRISE (N=44)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Cerebral artery occlusion (Nervous system disorders) | 1 (1)
Cerebral artery thrombosis (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arterial thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CODMAN ENTERPRISE (N=44)
Headache (Nervous system disorders) | 8 (8)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Urinary retention (Renal and urinary disorders) | 2 (4)
Vascular access complication (Injury, poisoning and procedural complications) | 3 (3)
Vasospasm (Vascular disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
Study was terminated due to a low rate of enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release and can embargo communications regarding trial results that is more than 60 days but less than or equal to 180 days from the time submitted to sponsor for review. No results that contain sponsor confidential information may be released without sponsor prior written consent.

DOCUMENTS (2):
  • Study Protocol (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT02532517/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT02532517/SAP_001.pdf